CLINICAL TRIAL: NCT05236673
Title: A Regulatory Requirement Non-interventional Study to Monitor the Safety and Effectiveness of Jardiance® (Empagliflozin, 10mg) in Korean Patients With Chronic Heart Failure (NYHA Class II-IV)
Brief Title: Jardiance® Post Marketing Surveillance (PMS) in Korean Patients With Chronic Heart Failure
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1245-0276
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — empagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who have started at first time on Jardiance®
  Interventions: Drug: JARDIANCE®

INTERVENTIONS:
Drug: JARDIANCE® — JARDIANCE® film-coated tablets 10mg
  Other Names: empagliflozin

SUMMARY:
The primary objective of this study is to monitor the safety profile of Jardiance® in Korean patient with chronic heart failure (New York Heart Association (NYHA) class II-IV) in a routine clinical setting.

ELIGIBILITY:
Inclusion criteria:

* Patients who have started at first time on Jardiance® in accordance with the approved label in Korea for heart failure (HF)
* Chronic heart failure (New York Heart Association (NYHA) class II-IV)
* Age ≥ 19 years at enrolment
* Patients who have signed on the data release consent form

Exclusion criteria:

* Patients with previous exposure to Jardiance®
* Known allergy or hypersensitivity to active ingredients empagliflozin or to any of the excipients
* Patients with type 1 diabetes or with prior history of diabetic ketoacidosis (DKA)
* Patient with renal impairment with estimated Glomerular Filtration Rate (eGFR) < 20 mL/min/1.73 m²
* Patients with rare hereditary conditions of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
* Patient who are pregnant or are nursing or who plan to become pregnant while in the trial
* Patients for whom empagliflozin is contraindicated according local label of Jardiance®

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with chronic heart failure (New York Heart Association (NYHA) class II-IV) in Korea.
Sampling Method: Non-Probability Sample
Enrollment: 610 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence rates of patients with adverse events | up to 24 weeks
  Adverse events will include: Adverse events, unexpected adverse events, unexpected adverse drug reaction, serious adverse events, serious adverse drug reaction, drug-related adverse events, non-serious adverse drug reaction, adverse event of special interest, adverse events leading to discontinuation.

SECONDARY OUTCOMES:
Occurrence of hospitalization for heart failure (first and recurrent) after 12 weeks of treatment from baseline | at week 12
Occurrence of hospitalization for heart failure (first and recurrent) after 24 weeks of treatment from baseline | at week 24
Occurrence of cardiovascular death after 12 weeks of treatment | at week 12
Occurrence of cardiovascular death after 24 weeks of treatment | at week 24
Changes from baseline in New York Heart Association (NYHA) functional class after 12 weeks of treatments | at baseline, at week 12
Changes from baseline in New York Heart Association (NYHA) functional class after 24 weeks of treatments | at baseline, at week 24
Changes in ejection fraction (EF) (if available) at 12 weeks compared to baseline | at baseline, at week 12
Changes in ejection fraction (EF) (if available) at 24 weeks compared to baseline | at baseline, at week 24
Changes in B-type Natriuretic Peptide (BNP) or N-terminal prohormone of brain natriuretic peptide (NT-proBNP) (if available) at 12 weeks compared to baseline | at baseline, at week 12
Changes in B-type Natriuretic Peptide (BNP) or N-terminal prohormone of brain natriuretic peptide (NT-proBNP) (if available) at 24 weeks compared to baseline | at baseline, at week 24
Changes in glycated hemoglobin (HbA1c) (if available in Type 2 Diabetes (T2D) patients) after 12 weeks of treatment | at baseline, at week 12
Changes in Fasting Plasma Glucose (FPG) (if available in Type 2 Diabetes (T2D) patients) after 12 weeks of treatment | at baseline, at week 12
Changes in glycated hemoglobin (HbA1c) (if available in Type 2 Diabetes (T2D) patients) after 24 weeks of treatment | at baseline, at week 24
Changes in Fasting Plasma Glucose (FPG) (if available in Type 2 Diabetes (T2D) patients) after 24 weeks of treatment | at baseline, at week 24
Change from baseline in estimated Glomerular Filtration Rate (eGFR) (if available) after 12 weeks of treatment | at baseline, at week 12
Change from baseline in estimated Glomerular Filtration Rate (eGFR) (if available) after 24 weeks of treatment | at baseline, at week 24
Change from baseline in body weight after 12 weeks of treatment | at baseline, at week 12
Change from baseline in body weight after 24 weeks of treatment | at baseline, at week 24
Change from baseline in blood pressure (systolic blood pressure (SBP), diastolic blood pressure (DBP)) after 12 weeks of treatment | at baseline, at week 12
Change from baseline in blood pressure (systolic blood pressure (SBP), diastolic blood pressure (DBP)) after 24 weeks of treatment | at baseline, at week 24
Investigator's overall effectiveness evaluation after 12 weeks of treatment | at week 12
  1. Improved: If determined as there is any effect of maintaining or improving disease related factors.
  2. Unchanged: If disease related factors have not been changed compared with before administration, and not determined as there is any effect of maintaining symptoms.
  3. Aggravated: If disease related factors are worse than before administration.
  4. Unassessable: If it cannot be determined due to insufficient information collected. (Even though there are any objective indicators present, it is possible to belong to this grade.) 'Improved' is assessed as "Effective", 'Unchanged' and 'Aggravated' are assessed as "Ineffective".
Investigator's overall effectiveness evaluation after 24 weeks of treatment | at week 24
  1. Improved: If determined as there is any effect of maintaining or improving disease related factors.
  2. Unchanged: If disease related factors have not been changed compared with before administration, and not determined as there is any effect of maintaining symptoms.
  3. Aggravated: If disease related factors are worse than before administration.
  4. Unassessable: If it cannot be determined due to insufficient information collected. (Even though there are any objective indicators present, it is possible to belong to this grade.) 'Improved' is assessed as "Effective", 'Unchanged' and 'Aggravated' are assessed as "Ineffective".

CONTACTS AND LOCATIONS:
Locations (21):
- South Korea (21):
  - Hallym University Medical Center, Anyang-si, Gyeonggi-do
  - Inje University Busan Paik Hospital, Busan
  - Inje University Haeundae Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Pusan National University Yangsan Hospital, Busan
  - Kangwon National University Hospital, Chuncheon-si, Gangwon-do
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Dongguk University Medical Center, Goyang-si, Gyeonggi-do
  - Inje University Ilsan Paik Hospital, Goyang-si, Gyeonggi-do
  - Chonnam National University Hospital), Gwangju
  - Jeonbuk National University Hospital, Jeonju-si, Jeollabuk-do
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - VHS Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul
  - Seoul National University Boramae Medical Center, Seoul
  - The Catholic University of Korea, Uijeongbu ST. Mary's Hospital, Uijeongbu-si, Gyeonggi-do

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com